CLINICAL TRIAL: NCT03599076
Title: Wearable Sensors for Quantitative Assessment of Motor Impairment in Huntington's Disease
Brief Title: Wearable Sensors for Quantitative Assessment of Motor Impairment in Huntington's Disease Huntington's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BioSensics (Industry)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: 1R44NS103648-01 (NIH)
Record Dates: First submitted 2018-06-27; First posted 2018-07-26 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Manifest HD
  Interventions: Other: HD Wear
- Premanifest HD
  Interventions: Other: HD Wear
- Control
  Interventions: Other: HD Wear

INTERVENTIONS:
Other: HD Wear — Wearable sensor system for monitoring Huntington's chorea during activities of daily living

SUMMARY:
The principal means of measuring motor impairment in Huntington disease (HD) is the Unified Huntington's Disease Rating Scale (UHDRS) total motor score, which is subjective, categorical, requires significant training to administer correctly, and only captures impairments in clinic. In this Direct to Phase II SBIR we will develop a wearable sensor system for objective, sensitive, and continuous assessment of Huntington's chorea during activities of daily living. The developed technology could be used clinically to detect changes in motor function in response to medications, or could be used scientifically to expedite and reduce the cost of early stage pharmaceutical clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* CAG expansion ≥ 36

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Huntington's Disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-09-25 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Chorea severity score | 12 months
  Remotely monitored chorea severity score based on movement data during activities of daily living

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No